CLINICAL TRIAL: NCT02032095
Title: The Desensitization Therapy With GB-0998 for Anti-donor Antibody-positive Recipients.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Japan Blood Products Organization (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B211-10
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: End Stage Renal Disease
Keywords: IVIG; Renal transplantation; desensitization
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GB-0998 (Experimental)
  Interventions: Drug: GB-0998

INTERVENTIONS:
Drug: GB-0998
  Other Names: Intravenous immunoglobulin (Venoglobulin IH)

SUMMARY:
It is intended to examine the safety and efficacy of desensitization therapy by GB-0998 (intravenous immunoglobulin) for the anti-donor antibody positive recipient in need of pre-transplant desensitization. Patients with positive FCXM-T after performing twice double filtration plasmapheresis (DFPP) therapy will receive GB-0998 1g/kg/day for four days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 4 or 5 on the CKD classification.
* Of the patients that wants a living-donor kidney transplant of ABO blood type compatible, patients with positive FCXM-T and negative CDC-T to the donor.
* Patients with positive FCXM-T after performing twice DFPP therapy

Exclusion Criteria:

* Patients who had taking to continue immunosuppressive drugs or steroids within 4 weeks before obtaining informed consent.
* Patients who had IVIG therapy, or plasmapheresis therapy within 12 weeks before to informed consent.
* Patients who had Rituximab within 6 month before to informed consent.
* Patients who have undergone splenectomy.
* Patients with severe hepatic disorder or severe heart disorder.
* Patients with receiving treatment of malignancy.
* Patients with high risk of thromboembolism.
* Patients with history of shock or hypersensitivity to GB-0998.
* Patients with hereditary fructose intolerance or IgA deficiency.
* Patients with pregnant or probably pregnant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-11; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Negative rate of FCXM-T after the fourth administration of GB-0998 | at 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Japan Blood Products Organization, Tokyo, Japan